CLINICAL TRIAL: NCT01322425
Title: Urocortins and Musculoskeletal Hyperalgesia
Brief Title: Effect of Temperature on Pain and Brown Adipose Activity in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1007M85352
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Fibromyalgia; Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The pathophysiology of pain related to fibromyalgia is not understood. This condition is difficult to diagnose and to treat. One clue may be that tender points (areas which hurt typical of fibromyalgia) are most densely located near the clavicles. This is also the area where brown fat is located in humans. Brown fat is typically used to maintain body temperature. Stress (such as cool temperature or special diets, i.e., high fat, low carbohydrate) appears to worsen the pain seen in fibromyalgia. We hypothesize that a mechanism for pain in this disease relates to activating brown fat through neural mechanisms. The nerves to brown fat also go into adjacent muscle and skin. So, when brown fat is turned on or increases in amount, collateral nerves may cause pain at the tender points.

The central hypothesis is that stress such as temperature or diet will activate brown fat. Patients with fibromyalgia will have greater activation or volume of brown fat. Neuralgia related to stress may be the etiology of the pain. If this hypothesis is proven, there are several drugs on the market that could be deployed to correct these patients' problems. Therefore, this project, if successful, will lead to clinical trials of these drugs in fibromyalgia patients.

DETAILED DESCRIPTION:
The pathophysiology of pain related to fibromyalgia is not understood. This condition is difficult to diagnose and to treat. One clue may be that tender points (areas which hurt typical of fibromyalgia) are most densely located near the clavicles. This is also the area where brown fat is located in humans. Brown fat is typically used to maintain body temperature. Stress (such as cool temperature or special diets, i.e., high fat, low carbohydrate) appears to worsen the pain seen in fibromyalgia. We hypothesize that a mechanism for pain in this disease relates to activating brown fat through neural mechanisms. The nerves to brown fat also go into adjacent muscle and skin. So, when brown fat is turned on or increases in amount, collateral nerves may cause pain at the tender points.

The central hypothesis is that stress such as temperature or diet will activate brown fat. Patients with fibromyalgia will have greater activation or volume of brown fat. Neuralgia related to stress may be the etiology of the pain. If this hypothesis is proven, there are several drugs on the market that could be deployed to correct these patients' problems. Therefore, this project, if successful, will lead to clinical trials of these drugs in fibromyalgia patients.

The initial study phase will involve five subjects - one healthy volunteer and four women with fibromyalgia. These five subjects will each have one visit that will include several hours in both the warm room and the cold room. Nociceptive flexion reflex (NFR) testing will be conducted while they are in each of the temperature-controlled rooms. We anticipate conducting the initial phase in the last two weeks of November 2010.

The main study project will entail three visits for each of 20 subjects (10 healthy control subjects and 10 women with fibromyalgia. No treatments are planned for this project.

Procedures include: a) screening interview, diagnostic interview, analog rating scales, and psychological and psychiatric rating scales; b) review of medical records if the diagnosis of fibromyalgia is not certain; c) pain will be measured by palpation at tender points and by measurement of biceps reflex that objectively measures amount of pain both before and after visits, d) Visit A will include a special diet for breakfast at 8 AM and resting at room temperature for 2.5 hours (both known to turn off brown fat) before receiving FDG (radioactive sugar) and a PET/CT scan to measure metabolism e) Visit B requires another diet and resting for 2.5 hours at ~62°F (both known to turn on brown fat) along with the PET/CT scan to measure metabolism and a structural MRI to examine brain structure and to measure volume of brown fat in chest; f) blood samples will be collected to measure stress hormones before and after each warm or cold period; g) pregnancy testing before PET/CT and MRI.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-50 years of age and premenopausal fibromyalgia or 30-50 years of age and premenopausal for healthy volunteers
* Healthy volunteer or diagnosis of fibromyalgia
* In follicular phase (Days 1-12) of menstrual cycle OR on contraceptives.
* Able to comply with study procedures.
* Capable of giving informed consent; consent obtained and form signed

Exclusion Criteria:

* Serious medical conditions (determined by investigator)
* Some medicines that affect brain metabolism (determined by investigator)
* Subjects who have participated in other studies with radioactivity may not be eligible depending on prior exposure
* BMI more than 35 kg/m2 (i.e. severe obesity)
* Pregnant or nursing females
* Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy or patients with fibromylgia
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Body temperature | 2 hours
  Body temperature was taken over a two hour interval at two different ambient temperatures.

CONTACTS AND LOCATIONS:
Overall Officials: Alice A. Larson, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States